CLINICAL TRIAL: NCT03695159
Title: The Perioperative Management of Anti-thrombotic Drug Registry
Acronym: CNCS
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Subhash Banerjee, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 012018-005
Record Dates: First submitted 2018-08-20; First posted 2018-10-03 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Surgery; Perioperative/Postoperative Complications
Keywords: anti-thrombotic drugs; cardiac intervention; Non-cardiac intervention
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate contemporary antiplatelet therapy management of patients referred for non-cardiac and cardiac surgical procedures while on chronic therapy with antiplatelet and/or anticoagulant drugs. These medications are routinely prescribed to patients following percutaneous coronary interventions (PCI), known diagnosis of atrial fibrillation, prosthetic heart valves, transcatheter aortic valve procedures, pulmonary embolism, deep vein thrombosis, peripheral artery revascularization procedures etc. This is a highly relevant and understudied clinical area with no randomized clinical trials or large-scale prospective evidence, except for bridging data with unfractionated heparin (UFH). Most recommendations and guidelines are based on consensus expert opinion. While post-PCI patients, especially those treated with coronary stents are placed on dual antiplatelet agents such as aspirin and P2Y12 blocking agents, performing surgery while on these agents increase the risk of hemorrhagic complications, discontinuation or interruption of dual antiplatelet therapy (DAPT) has been associated with adverse ischemic outcomes secondary to myocardial infarction (MI) and stent thrombosis (ST). Moreover, there is only no clear consensus regarding continuation of aspirin perioperatively in these patients. As in the case of PCI, similar arguments for juxtaposed risks (thrombosis vs. bleeding) can be made for a myriad of clinical situations where chronic (≥45 days) use antiplatelet and anticoagulant medication (together referred to as antithrombotic drugs) are indicated. In addition, there are many procedures and surgeries with different bleeding and ischemic risks that cannot be studies through dedicated randomized studies and a registry collection of such information could provide valuable guidance to providers and patients worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with antiplatelet and/or anticoagulant medications for ≥45 days prior to the date of NCS.
* Patients with planned, urgent or emergent cardiac or non-cardiac surgery or procedure (CNCS)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on chronic antiplatelet and anticoagulant therapies and undergo a cardiac and non-cardiac surgeries and procedures (CNCS)
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes (Net Adverse Cardiovascular events (%)) | time of study reporting initiation (14 days prior to CNCS) to end of study (30 days post-CNCS).
  A composite of Death, Non-Fatal MI, Ischemic Stroke, Need for Urgent Coronary Revascularization, and Bleeding (defined by Bleeding Associated Research Consortium- BARC)

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Study Chair — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - North Texas VA Health Care System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidbuchel H, Verhamme P, Alings M, Antz M, Hacke W, Oldgren J, Sinnaeve P, Camm AJ, Kirchhof P; European Heart Rhythm Association. European Heart Rhythm Association Practical Guide on the use of new oral anticoagulants in patients with non-valvular atrial fibrillation. Europace. 2013 May;15(5):625-51. doi: 10.1093/europace/eut083. PMID 23625942
- [Background] Beyer-Westendorf J, Gelbricht V, Forster K, Ebertz F, Kohler C, Werth S, Kuhlisch E, Stange T, Thieme C, Daschkow K, Weiss N. Peri-interventional management of novel oral anticoagulants in daily care: results from the prospective Dresden NOAC registry. Eur Heart J. 2014 Jul 21;35(28):1888-96. doi: 10.1093/eurheartj/eht557. Epub 2014 Jan 6. PMID 24394381
- [Background] Douketis JD, Spyropoulos AC, Kaatz S, Becker RC, Caprini JA, Dunn AS, Garcia DA, Jacobson A, Jaffer AK, Kong DF, Schulman S, Turpie AG, Hasselblad V, Ortel TL; BRIDGE Investigators. Perioperative Bridging Anticoagulation in Patients with Atrial Fibrillation. N Engl J Med. 2015 Aug 27;373(9):823-33. doi: 10.1056/NEJMoa1501035. Epub 2015 Jun 22. PMID 26095867
- [Background] Tsimikas S. Drug-eluting stents and late adverse clinical outcomes lessons learned, lessons awaited. J Am Coll Cardiol. 2006 May 16;47(10):2112-5. doi: 10.1016/j.jacc.2006.03.019. Epub 2006 Apr 4. No abstract available. PMID 16697332
- [Background] Cruden NL, Harding SA, Flapan AD, Graham C, Wild SH, Slack R, Pell JP, Newby DE; Scottish Coronary Revascularisation Register Steering Committee. Previous coronary stent implantation and cardiac events in patients undergoing noncardiac surgery. Circ Cardiovasc Interv. 2010 Jun 1;3(3):236-42. doi: 10.1161/CIRCINTERVENTIONS.109.934703. Epub 2010 May 4. PMID 20442357